CLINICAL TRIAL: NCT03429491
Title: Novel Nutrition Solutions in Elderly at Risk of Sarcopenia: LC n-3 PUFA and Leucine Combinations
Brief Title: Novel Nutrition Solutions for Sarcopenia
Acronym: NUTRIMAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College Dublin (Other)
Responsible Party: Principal Investigator, Prof Helen M Roche, Professor Helen Roche, University College Dublin
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: NUTRIMAL-3; 14/F/822 (Other Grant/Funding Number: Department of Agriculture and Marine)
Record Dates: First submitted 2018-02-03; First posted 2018-02-12 (Actual); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Sarcopenia
MeSH Terms: conditions — Sarcopenia | interventions — P3H1 protein, human

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Protein-free, LC n-3 PUFA-free juice based supplement
  Interventions: Dietary Supplement: Placebo
- Leucine-enriched protein (Experimental): Juice based supplement containing leucine-enriched protein
  Interventions: Dietary Supplement: Leucine-enriched protein
- Leucine-enriched protein + LC n-3 PUFA (Experimental): Juice based supplement containing leucine-enriched protein and LC n-3 PUFA
  Interventions: Dietary Supplement: Leucine-enriched protein; Dietary Supplement: LC n-3 PUFA

INTERVENTIONS:
Dietary Supplement: Placebo — Protein-free, LC n-3 PUFA-free juice based supplement
  Arms: Placebo
Dietary Supplement: Leucine-enriched protein — Leucine-enriched whey protein
  Arms: Leucine-enriched protein; Leucine-enriched protein + LC n-3 PUFA
Dietary Supplement: LC n-3 PUFA — LC n-3 PUFA
  Arms: Leucine-enriched protein + LC n-3 PUFA

SUMMARY:
This study will examine the effect of leucine-enriched protein supplementation, alone and in combination with long chain n-3 polyunsaturated fatty acids (LC n-3 PUFA), on muscle mass and function in older adults at risk of sarcopenia.

The investigators hypothesize that LC n-3 PUFA supplementation will further enhance the efficacy of the leucine-enriched protein.

DETAILED DESCRIPTION:
The progressive loss of skeletal muscle mass and function with advancing age, termed sarcopenia, contributes substantially to disability, physical dependence, and mortality among older adults. Aging is associated with an attenuated muscle protein synthetic response to the ingestion of small to moderate protein doses compared to younger persons. Several studies have reported that the acute, postprandial muscle protein synthesis (MPS) response to a suboptimal protein dose is enhanced when the leucine content of the protein bolus is increased. This indicates that supplementing the lower-protein daily meals (i.e., breakfast and lunch) with leucine may represent a practical strategy to augment the MPS response to these meals and, subsequently, attenuate sarcopenic muscle mass loss over time. In addition, LC n-3 PUFA supplementation has been shown to enhance the MPS response to amino acid infusion older adults suggesting that combined leucine and LC n-3 PUFA supplementation be particularly effective for improving daily MPS, muscle mass and function in older adults.

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥65 y
* Sex: males and females
* Low muscle mass (assessed via bioelectrical impedance analysis using cut-offs from Janssen, 2004) and/or low handgrip strength (< 30 kg men, <20kg women)

Exclusion Criteria:

* BMI >35 kg/m2
* Cancer - malignancy in the past 5 years
* Multiple Sclerosis, Parkinsons Disease
* Chronic kidney disease
* Liver failure
* Diabetes
* Conditions that will affect ability to consume, digest and/or absorb the study drink (i.e. cows milk protein allergy, inflammatory bowel disease)
* Smokers
* Cognitive function < 21 on Mini-Mental State Examination
* Excess alcohol intake
* Regular resistance training
* Total walking incapacity
* Musculoskeletal or neuromuscular impairments that could interfere with strength testing
* Medications interfering with muscle metabolism
* Adherence to a high energy or high protein diet three months before starting and during the study. Use of protein containing or amino acid containing nutritional supplements three months before starting and during the study.
* High consumers of oily fish.
* Weight change > 3 kg past 3 months

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 108 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-12-21 (Actual); Study Completion 2018-12-21 (Actual)

PRIMARY OUTCOMES:
Appendicular skeletal muscle mass | 6 months
  Assessed via dual energy x-ray absorptiometry

SECONDARY OUTCOMES:
Isometric knee extension strength | 6 months
  Maximal voluntary contraction
Physical performance | 6 months
  Short physical performance battery, single leg stand, timed up and go
Metabolomics | 6 months
  Assessed using nuclear magnetic resonance (NMR) spectroscopy
Transcriptomics | 6 months
  Assessed via RNA Sequencing
Thigh muscle mass | 6 months
  Assessed in dominant leg via MRI in sub cohort (n=39)
Muscle protein synthesis | 6 months
  Measured as fractional synthetic rate (%/day) over a 3-d period at baseline and end of study

CONTACTS AND LOCATIONS:
Overall Officials: Helen Roche, PhD, Principal Investigator — University College Dublin
Locations (1):
- University College Dublin, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Murphy CH, Flanagan EM, De Vito G, Susta D, Mitchelson KAJ, de Marco Castro E, Senden JMG, Goessens JPB, Miklosz A, Chabowski A, Segurado R, Corish CA, McCarthy SN, Egan B, van Loon LJC, Roche HM. Does supplementation with leucine-enriched protein alone and in combination with fish-oil-derived n-3 PUFA affect muscle mass, strength, physical performance, and muscle protein synthesis in well-nourished older adults? A randomized, double-blind, placebo-controlled trial. Am J Clin Nutr. 2021 Jun 1;113(6):1411-1427. doi: 10.1093/ajcn/nqaa449. PMID 33871558